CLINICAL TRIAL: NCT02620189
Title: A Study to Investigate the Role of IL-17 and Th17 Pathway Activation in RA Patients With Inadequate Response to Anti-TNFα Therapies
Brief Title: Th17 Responses Evaluated in RA Patients on Inhibitors of TNFα
Acronym: THERAPIST
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 009745
Record Dates: First submitted 2015-10-12; First posted 2015-12-02 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab; Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Synovial tissue
  * RNA extraction on peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anti-TNF Biologics Therapy
  Other Names: Etanercept (Enbrel); Adalimumab (Humira); Certolizumab Pegol(Cimzia)

SUMMARY:
Preliminary data suggest that up-regulation of Interleukin -17 (IL-17) and the T-helper 17 (Th17) pathway occurs in rheumatoid arthritis (RA) patients on anti-Tumour Necrosis Factor (TNF) therapy who demonstrated an incomplete clinical response. A deeper understanding of this is required in order to determine whether IL-17 or the Th17 pathway is a valid target for intervention in this population to improve response outcome.

The study objective is to observe biologic naïve RA subjects on anti-TNF therapies and take measurements of peripheral blood and synovial tissue to assess differences in the IL-17 and Th17 pathways between responders and non-responders. The aim of the study is to test if increased Th17 pathway activity is present in subjects who do not respond clinically to anti-TNF therapy.

Clinical assessments, synovial bio-markers and ultrasound will be used as determinants of clinical response. The study may identify disease characteristics that determine which subjects may be more likely to respond to anti-TNF therapy, or those who may require either a different treatment option, or additional pathway inhibition in addition to TNF, in order to achieve clinical response.

DETAILED DESCRIPTION:
The study aims to recruit 50 participants in total to this study. Potential candidate for this research include those that have active rheumatoid arthritis (RA) with the symptoms, and current medication status that qualify for anti-TNFα therapy. This is the treatment plan patients will be placed on regardless of whether or not they are taking part in the study; however, within the research environment, information will be gathered that may be able to help better understand the levels of response to anti-TNF treatment and why this differs between people. Participants will be asked to provide blood and urine samples as part of the research. Pieces of genetic material called ribonucleic acid (RNA) will be extracted from the study specific blood samples (and synovial tissue from patients that are part of the biopsy sub-study) provided by participants. This material will be analysed to reveal information about what genes are 'active' in the joint environment during anti-TNF treatment period. This information can tell us what proteins might be involved in the inflammation of affected joints and might also be able to predict what type of response patients will experience in response to different treatments. The analysis of research samples from this study will provide new information on the mechanisms for response/non-response to anti-TNF therapy.

Optional Biopsy sub-study A number of participants that have consented to the main study will be invited to take part in the optional biopsy sub-study. This will involve taking a biopsy of one of the affected joints via an ultrasound guided procedure. The procedure is minimally invasive and has good safety and tolerability with participants. The procedure is performed under local anaesthetic and removes tiny pieces of inflamed tissue (synovial tissue) from the lining of the joint using a needle under the guidance of an ultrasound scanner. This sub-study will collect tissue from affected joints to help answer the research questions in this study

Optional DNA genetic sampling Participants are also invited to take part in the optional DNA genetic sampling and are asked to contribute DNA samples for this study. The purpose of this optional part of the research study is to help understand how anti-TNF therapies work, and how they may cause side effects, to further understand rheumatoid arthritis, and to understand why some people respond to anti-TNF therapy while others do not. Genetic (genotyping) testing refers to patient sample being used for genetic research. This is the study of DNA and how it determines our traits. DNA research can also explain why some people respond well to their medications and others do not and can also provide reasons as to why some people develop some diseases and others do not. Samples from participants that have consented to the optional DNA genetic sampling will also be used for a type of genetic research called epigenetics. This is the study of chemical modifications of DNA that occur over time, without a change in DNA sequence. These modifications control the way cells produce proteins and respond to the environment. Epigenetics research is not a test to diagnose a person for a genetic disease or to determine whether a person may have a risk of developing a genetic disease. It is only used to understand prevailing disease and how drugs may work in different groups of people. In epigenetic testing, DNA samples from participants will be analysed to determine how this may influence response to anti-TNF therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age
2. An RA diagnosis as defined by the 2010 revised EULAR/ACR classification criteria.
3. Subjects who fulfil the NICE guidelines for Biologic therapy as their first line treatment following failure of standard disease modifying anti-rheumatic therapy.
4. Subjects may be on cDMARDs (or MTX monotherapy) one of which must be MTX. Participants should be receiving MTX for at least 2 months at a stable dose of 7.5-25 mg/week before Week 0 visit.
5. Subjects may be on oral steroids (prednisone ≤10 mg/day, or equivalent corticosteroid) with a stable dose for the 4 weeks prior to Week 0 visit.
6. Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) for the duration of the study.
7. Participants must be able to adhere to the study visit schedule.
8. The participant must be capable of giving informed consent and the consent must be obtained prior to any screening procedures.
9. Must have a chest X-ray within 6 months prior to commencement of anti-TNF therapy with no evidence of malignancy, infection or fibrosis.

Exclusion Criteria:

Participants will be excluded from this study for any of the following reasons:

1. Women who are pregnant or breast feeding.
2. Previous use of Rheumatoid Arthritis anti-TNF biologics, or ANY other type of biologic therapy or Investigational Medicinal Product.
3. Treatment with any other therapeutic agent targeted at reducing TNF within 3 months of screening.
4. Serious infections (such as pneumonia or pyelonephritis) in the previous 3 months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
5. Known HIV, Hepatitis B, or Hepatitis C infection.
6. Have active TB or have evidence of latent TB (old or latent TB on chest x-ray, without adequate therapy for TB initiated prior to first dose of study drug). Participants with a current close contact with an individual with active TB and participants who have completed treatment for active TB within the previous 2 years are explicitly excluded from the trial. Participants with a household member who has a history of active pulmonary TB should have had a thorough evaluation for TB prior to study enrolment as recommended by a local infectious disease specialist or published local guidelines of TB control agencies.
7. Presence of a transplanted organ (with the exception of a corneal transplant >3 months prior to screening).
8. Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
9. History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly.
10. Known recent substance abuse (drug or alcohol).
11. Poor tolerability of venepuncture required blood sampling during the study period.
12. Planning to have surgery for RA or other significant surgery during the period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who fulfil the NICE guidelines for biologic anti-TNF therapy as their first line treatment following failure of standard disease modifying anti-rheumatic therapy will be recruited from various secondary care settings at a number of centres throughout the UK.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Measure change in clinical response using Disease Activity Score DAS28 (C-Reactive Protein) at week 24 compared to baseline | Baseline and week 24
  Change in clinical response using Disease Activity Score DAS28 (C-Reactive Protein) at week 24 compared to baseline

SECONDARY OUTCOMES:
Change in Interleukin (IL)-17/T helper (Th)17 pathway activity in responders and non-responders to anti-Tumour Necrosis Factor (TNF) therapy | Baseline and week 24
  Correlation of the change in IL-17/Th17 pathway activity and ultrasound assessment of synovitis by grey-scale ultrasound and power Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Costantino Pitzalis, MD PhD FRCP, Study Chair — Queen Mary University of London
Locations (8):
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Barts Health NHS Trust, Experimental Medicine & Rheumatology, Mile End Hospital, London
  - Barts Health NHS Trust,Department of Rheumatology,Whipps Cross University Hospital, London
  - University College London Hospitals NHS Foundation Trust, Rheumatology Department, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, The Kellgren Centre for Rheumatology, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Royal Victoria Infirmary, Newcastle
  - Oxford University Hospitals NHS Trust, Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences, Oxford